CLINICAL TRIAL: NCT05099796
Title: Comparison of Caudal Versus Transforaminal Epidural Steroid Injection in Post-lumbar Surgery Syndrome After Single-level Discectomy: A Prospective, Randomized Clinical Trial
Brief Title: Epidural Steroid Injections in Post-lumbar Surgery Syndrome After Single-level Discectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09.2014.0085
Record Dates: First submitted 2021-10-11; First posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Failed Back Surgery Syndrome; Low Back Pain; Radiculopathy; Epidural Fibrosis
Keywords: Failed back surgery syndrome, epidural steroid injections
MeSH Terms: conditions — Failed Back Surgery Syndrome; Low Back Pain; Radiculopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Transforaminal epidural steroid injection (TESI) group (Active Comparator): This procedure was applied only once.
  1 to 2 cc of the contrast agent (300 mg/50 mL iohexol) was given and the distribution pattern was visualized. Once the epidural distribution of the contrast agent was confirmed without vascular flow, a mixture of 40 mg (1mL) of triamcinolone acetonide, 2 cc of physiological saline, and 2 cc (0.5%) of bupivacaine was injected.
  Interventions: Procedure: Transforaminal epidural steroid injection
- Caudal epidural steroid injection (CESI) group (Active Comparator): This procedure was applied only once
  1 to 2 cc of the contrast agent (300 mg/50 mL iohexol) was given and the distribution pattern was visualized which showed bilateral L5-S3 distribution without vascular flow. A mixture of 40 mg (1mL) of triamcinolone acetonide, 7 cc of physiological saline, and 2 cc (0.5%) of bupivacaine was injected. A total of 10 cc mixture was used for CESI.
  Interventions: Procedure: Caudal epidural steroid injection

INTERVENTIONS:
Procedure: Transforaminal epidural steroid injection
  Arms: Transforaminal epidural steroid injection (TESI) group
Procedure: Caudal epidural steroid injection
  Arms: Caudal epidural steroid injection (CESI) group

SUMMARY:
62 patients with postlumbar surgery syndrome were randomized and divided into two groups. Transforaminal epidural steroid injection (TFESI) was applied to the TFESI group (n=31), and caudal epidural steroid injection (CESI) was applied to the CESI group (n=31). The age of the patients involved in this study ranged from 18 years old to 65 years old

DETAILED DESCRIPTION:
Patients with low back and radicular pain related to epidural fibrosis following single-level lumbar discectomy were included. The patients were randomly divided into two groups as the CESI group and TFESI group. Transforaminal epidural steroid injection was applied to the TFESI group (n=31), and caudal epidural steroid injection was applied to the CESI group (n=31). All patients were assessed before the procedure (baseline) and at 1 hour, three weeks, and three months after the procedure using the Numerical Rating Scale (NRS) and at baseline and three weeks and three months using the modified Oswestry Disability Index (mODI). Treatment success was defined as ≥50% decrease in the NRS scores compared to baseline

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Previous single-level, open, non-fusion discectomy for L4-5 or L5-S1 lumbar disc herniation within the past six months
* Having epidural fibrosis involving the L4, L5 or S1 nerve root on magnetic resonance imaging
* Having low back and leg pain for at least six months and unresponsive to conservative therapies
* A Numerical Rating Scale score of ≥4
* Having a single-level epidural fibrosis in the operated level and side as assessed by contrast-enhanced spinal magnetic resonance imaging

Exclusion Criteria:

* Having a multi-level epidural fibrosis
* Previous surgery for multi-level disc herniation
* Previous lumbar fusion surgery
* Having recurrent disc hernia
* Having sacroiliac/facet joint pain
* Having lumbar spinal stenosis, spondylolysis, spondylolisthesis, or scoliosis
* History of epidural steroid injection within the past six months
* Having bleeding diathesis
* Presence of systemic or local infections
* Pregnancy
* Known hypersensitivity to the injectates to be applied

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-01-05 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-05-11 (Actual)

PRIMARY OUTCOMES:
Change in pain severity | All patients were assessed from baseline to each checkpoint (at 1 hour, three weeks, and three months after the procedure)
  Numerical Rating Scale (NRS) is a scale for assessing the severity of pain. The numerical rating scale ranges from 0 to 10, with 0 being "no pain" and 10 being "worst pain imaginable". The patient chooses the most appropriate number describing the severity of pain (oral version).
Change in disability score | All patients were assessed from baseline to each checkpoint (at 1 hour, three weeks, and three months after the procedure)
  Modified Oswestry Disability Index (MODI) is a 10-question questionnaire assessing disability in low back pain. Each question has 6 options. The lowest score for each question is zero and the highest score is 5. High score is associated with increased disability.

CONTACTS AND LOCATIONS:
Overall Officials: Savas Sencan, Assoc. Prof., Study Director — Marmara University Pendik Training and Research Hospital
Locations (1):
- Marmara University Pendik Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided